CLINICAL TRIAL: NCT02390193
Title: Effect of Hemodialysis on Upper Airways Collapsibility in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário de Anapolis (Other)
Collaborators: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Luis Vicente Franco de Oliveira, PhD, Centro Universitário de Anapolis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 368856/2010
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Chronic kidney disease; Dialysis; Sleep; Pulmonary function; Polysomnography; Upper airway
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hemodialysis (Experimental): Chronic kidney disease patients undergoing hemodialysis will be recruited consecutively and screened for eligibility using a standardised protocol.
  Interventions: Procedure: Hemodialysis

INTERVENTIONS:
Procedure: Hemodialysis — Daytime haemodialysis was standardised. It was performed 3 times per week, with a 4-h session duration, 250-mL/min blood flow, and 500-mL/min dialysate flow, using bicarbonate buffered dialysate with 1.25 mmol/L ionised calcium concentration, dialysate temperature of 36.5°C.
  The ultrafiltration amount for each haemodialysis session was decided by individual dry weight, which was fixed during the trial. In addition, the patients were not permitted to change their medication or start new drugs, especially antiplatelet agents, angiotensin-converting enzyme inhibitors, angiotensin II receptor antagonists, calcium-channel blockers, and β-blockers.
  The patients who required a change in medication for medical reasons were subsequently excluded from the study.

SUMMARY:
Introduction: Currently, chronic kidney disease (CKD) is one of the most serious public health problems, becoming a global epidemic. It is also known that the amount of displacement of overnight rostral fluid, from the lower limbs, is related to increased neck circumference and severity of obstructive sleep apnea (OSA) in patients with end-stage renal disease. Method / Design: A clinical trial study aiming to assess the degree of collapsibility of the upper airway in patients with CKD undergoing hemodialysis has been proposed. The test of the negative expiratory pressure and nocturnal polysomnography will be performed before and after the hemodialysis session. Discussion: The incidence of CKD has increased, due to the increased number of cases of diabetes mellitus and hypertension. Our hypothesis is that the weight gain due to volume overload, observed in the interdialytic period, will exert a negative influence on the degree of collapsibility of the upper airways predispose to OSA in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients aged 18 to 80 years;
* chronic kidney failure;
* candidate for kidney transplant with indication for dialysis;
* cognitive level sufficient for understanding the procedures and following the instructions;
* absence of dementia or treatment-refractory psychiatric diseases leading to an inability to provide informed consent.
* and agreement to participate by signing a statement of informed consent.

Exclusion Criteria:

* craniofacial abnormalities;
* undergoing active treatment of sleep apnea;
* active malignancy;
* active alcohol and/or drug abuse;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2015-01-02; Primary Completion 2018-05-02 (Actual); Study Completion 2020-12-03 (Estimated)

PRIMARY OUTCOMES:
Collapsibility of the upper airway. | 06 months
  Degree of upper airway collapsibility through the negative expiratory pressure test in patients with chronic kidney disease on hemodialysis.

SECONDARY OUTCOMES:
Prevalence and severity of sleep disorders | 06 months
  To assess the effects of dialysis on sleep parameters and determine the prevalence and severity of sleep disorders.
Change in pulmonary function. | 06 months
  Lung function tests will be performed during the day, with the patient seated in a comfortable position. For such, the KoKo PFT Spirometer System version 4.11 (nSpire Health, Inc, Louisville, CO, USA) will be used in accordance with the guidelines for the execution of lung function tests established by the Brazilian Society of Pneumology and European Respiratory Society.

CONTACTS AND LOCATIONS:
Overall Officials: Luis VF Oliveira, PhD, Study Chair — Centro Universitário de Anápolis - UniEVANGÉLICA
Locations (1):
- Centro Universitário de Anápolis - UniEVANGÉLICA, Anápolis, Goiás, Brazil